CLINICAL TRIAL: NCT05062434
Title: Improving Safety of Cardiovascular Implantable Electronic Devices in Veterans (CDA 21-057)
Brief Title: An Intervention to Impact Cardiovascular Implantable Electronic Device Lead Models Implanted in Veterans
Acronym: Veteran CIEDs
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: CDX 21-007; 1IK2HX003357-01A1 (NIH)
Record Dates: First submitted 2021-09-09; First posted 2021-09-30 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Patient Safety
Keywords: Defibrillators, Implantable; Pacemaker, Artificial

STUDY DESIGN:
Intervention Model Description: This is a pilot study for cardiac electrophysiologists at 3 Veterans Integrated Service Networks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention Arm (Experimental): VA cardiac electrophysiologists receiving the intervention
  Interventions: Other: Academic detailing and audit and feedback intervention

INTERVENTIONS:
Other: Academic detailing and audit and feedback intervention — An academic detailing and audit and feedback intervention will be presented to VA cardiac electrophysiologists, and will include quantitative data about the individual physician's facilities cardiovascular implantable electronic device lead implants and national data on lead implants over the past year.

SUMMARY:
This study will evaluate if an intervention using academic detailing and audit and feedback impacts the specific pacemaker or implantable cardioverter-defibrillator (ICD) lead models implanted in Veterans.

DETAILED DESCRIPTION:
This study will identify Department of Veterans Affairs (VA)-based cardiac electrophysiologists at three Veterans Integrated Service Networks (VISNs). Each cardiac electrophysiologist will participate in a videoconference during which time an academic detailing and audit and feedback intervention will be implemented, which will include details and recommendations about lead selection for implantation, based on cardiovascular implantable electronic device (CIED: pacemaker and implantable cardioverter-defibrillator [ICD]) lead-specific failure rates for lead models currently available in clinical practice. The cardiac electrophysiologist will also be presented with quantitative data about the individual physician's facility's implants and national data on implants over the past year. These data will be shared in advance, with time for questions and discussion. The electrophysiologist will be asked if anything can be done to facilitate selection of CIED lead models with the statistically and clinically significantly lower failure rates.

Then, over the subsequent 3 months, a quantitative evaluation of the CIED lead models implanted will be evaluated, comparing changes in lead model selection among the electrophysiologists receiving the intervention to a control group of all VA cardiac electrophysiologists who do not receive the intervention. Subsequently, semi-structured interviews will be conducted to assess reasons for changes, or lack thereof, in CIED lead model selection - including barriers and facilitators. Finally, quantitative data will be included to each of the cardiac electrophysiologists, with additional feedback.

ELIGIBILITY:
Inclusion Criteria:

* Department of Veterans Affairs-based cardiac electrophysiologists who implant cardiovascular implantable electronic devices at three Veterans Integrated Service Networks (VISNs)

Exclusion Criteria:

* Not willing to participate in the study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03-02 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of cardiovascular implantable electronic device leads that are of the lead model with the lowest failure rate | 3 months
  This outcome will be the proportion of cardiovascular implantable electronic device leads implanted in the 3 months post-intervention that are of the lead model with the lowest failure rate. The failure rates for the lead models will be available from VA data.

CONTACTS AND LOCATIONS:
Overall Officials: Sanket Shishir Dhruva, MD MHS, Principal Investigator — San Francisco VA Medical Center, San Francisco, CA
Locations (1):
- San Francisco VA Medical Center, San Francisco, CA, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No